CLINICAL TRIAL: NCT05147714
Title: The Relationship on The Surgical Pleth Index Values Observed at The End of The Surgical Procedure With Postoperative Pain Score and Analgesia Consumption
Brief Title: The Relationship Of The Surgical Pleth Index Values With Postoperative Pain Score And Analgesia Consumption
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dilek Hundur, Dr, Istanbul University
Other Study IDs: 2018/936
Record Dates: First submitted 2021-12-06; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Acute Pain; Analgesia
Keywords: Surgical pleth index; Craniotomy
MeSH Terms: conditions — Acute Pain; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Surgical Pleth Index (SPI) — SPI data were recorded at one-minute intervals during the last five minutes (6 times in total) until the entropy value reached 60

SUMMARY:
Postoperative pain management has an important role in anesthesia practice. In order to ensure postoperative patient comfort, postoperative rehabilitation should start early and be managed effectively1. It is known that if adequate analgesia is not provided before the patient wakes up, the severity of pain and the total opioid consumption increases. This increased opioid use causes complications such as nausea, vomiting, constipation, increased sleepiness and respiratory depression2. For this reason, the provision of adequate analgesia before the patient is awakened from general anesthesia has an important place in the process. Measurement of pain has different characteristics in patients under sedation or general anesthesia compared to conscious patients. However, since it is not possible for the patient to define pain under general anesthesia, different measurement and evaluation methods are needed. In order to monitor the intraoperative balance between nociception and antinociception, several non-invasive methods with different physiological approaches have been researched and made available for use in the last decade. The aim of these methods is individualize the intraoperative and postoperative opioid dose3. In this context, it has been suggested that the Surgical Pleth Index (SPI) method can be used in the evaluation of the analgesic component of anesthesia.

DETAILED DESCRIPTION:
After arrival in the operating room, patients were monitored with electrocardiogram (ECG), non-invasive arterial pressure measurement, pulse oximetry, neuromuscular monitoring (GE Datex, Ohmeda TOF module), entropy (GE Datex, Ohmeda Entropy Module) and SPI. Intravenous midazolam (0.03-0.05 mg/kg), fentanyl (1mcg/kg) were used before induction of anaesthesia. For anesthetic induction, propofol was administered until the entropy value fell below 60, followed by rocuronium was performed intravenous 0.6mg/kg. Patients were intubated with endotracheal tube than the mechanical ventilation was initiated with a mixture of O2 and air with FiO2 0.5 and adjusted to maintain end-tidal CO2 pressure of 35 and 40 mmHg. Intravenous propofol and remifentanil infusion were used for anesthesia maintenance and entropy was maintained below 60. Furthermore, SPI was maintained below 50.

Tenoxicam 20 mg, paracetamol 1 g and 0.5 mg/kg tramadol intravenously were administered 30 minutes before the end of the surgery to each patient who had no contraindications. After the last suture, the anesthetic agents were stopped and was considered the end of the surgery. Then SPI data were recorded at one-minute intervals during the last five minutes (6 times in total) until the entropy value reached 60. Patients who has cooperation were extubated and taken to the recovery room. The first time that the patients cooperated in the recovery room was considered as the zeroth minute. During the postoperative observation, the patient's pain score was questioned using the Numeric Rating Scale (NRS) every five minutes. If NRS≥4, intravenous tramadol 10 mg (100 mg as the maximum dose) was administered to the patient. The patient was followed in the recovery room for 30 minutes and until NRS <4. However, if NRS≥4 was still present at the end of the observation period, an additional 2 mg dose of morphine was administered. The maximum dose of morphine was determined as 0.1mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* ASA physical status I-III
* Who received craniotomy and intracranial mass excision

Exclusion Criteria:

* Diagnosed diabetic neuropathy
* Using pacemaker
* Needing vasoactive agent during the observation
* Using ketamine
* Using agents such as beta-blockers, beta-agonists, sympatholytic agents, atropine, neostigmine that will affect the sympatho-vagal balance during the observation period
* The patients who could not provide sufficient cooperation for scoring were not included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 65 years with ASA physical status I-III who received craniotomy and intracranial mass excision in the ITF Neurosurgery Clinic were enrolled in the study after providing written informed consent
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Acute Postoperative Pain | Postoperative 30 minutes
  During the postoperative observation, the patient's pain score was questioned using the Numeric Rating Scale (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Mukadder Orhan Sungur, Prof., Study Director — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No